CLINICAL TRIAL: NCT04977544
Title: A Randomized Controlled Study of Virtual Reality Exposure Therapy in the Intensive Treatment of Social Anxiety Disorder
Brief Title: Virtual Reality Exposure Therapy in the Intensive Treatment of Social Anxiety Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019232
Record Dates: First submitted 2021-06-20; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-06

CONDITIONS: Phobia
Keywords: phobia; VR
MeSH Terms: conditions — Phobic Disorders | interventions — Sertraline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drug only (Active Comparator): Sertraline was given as a single drug, with an initial dose of 50 mg/d, and gradually increased to the maximum dose of 200 mg/d after 2 weeks. The treating physician will determine the specific dose adjustment according to the patient's condition.
  Interventions: Drug: Sertraline
- vert combine with drug (Experimental): On the basis of sertraline drug treatment, phobia patients were given 2d/times from the 5th week, each 35-45min VR exposure treatment, 15 times as a course of treatment.
  Interventions: Device: vert; Drug: Sertraline

INTERVENTIONS:
Device: vert — On the basis of sertraline drug treatment, phobia patients were given 2d/times from the 5th week, each 35-45min VR exposure treatment, 15 times as a course of treatment.
  Arms: vert combine with drug
Drug: Sertraline — Sertraline was given as a single drug, with an initial dose of 50 mg/d, and gradually increased to the maximum dose of 200 mg/d after 2 weeks. The treating physician will determine the specific dose adjustment according to the patient's condition.

SUMMARY:
To explore the efficacy of drugs combined with virtual reality exposure therapy in the treatment of phobias compared with single drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for phobias in DSM-IV.
* Age from 18 to 45 years old.
* Graduated from junior high school or above.
* No serious physical disease, no serious visual impairment, and no family history of mental illness.

Exclusion Criteria:

* Exclude other psychiatric diagnosis and treatment history.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
the level of anxiety | 3 months
  the score of Hamilton anxiety scale, the minimum and maximum values are 0 and 56, and higher scores mean a worse outcome.
heart rate of the patients | 3 months
  take the heart rate as a biomarker of fear, the faster heart rate means the participate is more afraid

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University Medical College, Yiwu, Zhejiang, China